CLINICAL TRIAL: NCT07157176
Title: Laughie Prescription on the Well-being, Happiness, and Posttraumatic Stress Level of Nursing Students Affected by the Earthquake in Türkiye: A Randomized Controlled Trial
Brief Title: Laughie Prescription on the Well-being, Happiness, and Posttraumatic Stress Level of Nursing Students Affected by the Earthquake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Collaborators: University of Derby (Other); Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Nilgun Kuru Alici, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: D69072; Hacettepe University (Registry Identifier: Hacettepe University); Hacettepe University (Other: Hacettepe University)
Record Dates: First submitted 2025-08-16; First posted 2025-09-05 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-02

CONDITIONS: Well Being; Happiness; Post Traumatic Stress Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Daily 3-Minute Laughter Practice (Laughie Prescription)"
  Interventions: Behavioral: Daily 3-Minute Laughter Practice (Laughie Prescription)
- No Intervention (No Intervention): Control group The control group will not take part in the Laughie Prescription

INTERVENTIONS:
Behavioral: Daily 3-Minute Laughter Practice (Laughie Prescription) — The intervention will consist of 3-minutes of laughter (joyful and natural laughter is recommended) per day. Each day participants will laugh for one minute in a group (virtual and/or actual) guided by a professional laughter practitioner who is not going to be involved in the analysis of the data. That laughter will be recorded. The recording (the "Laughie") will then be prescribed for participants to laugh with (with others - family, friends, colleagues, or alone) twice a day. This will result in 3 minutes of laughter per day (the first in a group, the second two prompted by the Laughie)
  Arms: Experimental group

SUMMARY:
This study aimed to evaluate the effect of the Laughie Prescription on Well-being, Happiness, and Postraumatic stress levels of nursing students affected by the earthquake in Türkiye. The study hypothesises that the Laughie Prescription would have a positive effect on well-being, happiness, and lowering post-traumatic stress level scores among nursing students affected by the earthquake in Türkiye. The CONSORT-SPI 18 Checklist for the reporting of randomised trials of social and psychological interventions was adhered to in the development of this protocol.

DETAILED DESCRIPTION:
Purpose: The aim of the research is to examine the effects of the Laughie Prescription: if it would have a positive effect on well-being, happiness, and post-traumatic stress level scores among nursing students affected by the earthquake in Türkiye.

Methods: The study will conduct with 60 (30 in the intervention group, and 30 in the control group) nursing students. The study population in the intervention group will apply the intervention three times a day for one week. No intervention will be offered to the control group.

Recruitment: Participants will be recruited from the School of Nursing at XX University, in Hatay Turkiye - recruitment will be voluntary Randomization: Participants will be randomly assigned to either the control or the intervention group through a block randomisation prompt, where the block size is 5, within the Qualtrics link at the time participants sign up to the study. Authors involved in the analysis of the data will be blinded to participants' group allocation.

Intervention: The intervention will consist of 3-minutes of laughter (joyful and natural laughter is recommended) per day. Each day participants will laugh for one minute in a group (virtual and/or actual) guided by a professional laughter practitioner who is not going to be involved in the analysis of the data. That laughter will be recorded. The recording (the "Laughie") will then be prescribed for participants to laugh with (with others - family, friends, colleagues, or alone) twice a day. This will result in 3 minutes of laughter per day (the first in a group, the second two prompted by the Laughie).

Data will be collected with a socio- demographic questionnaire, and Well-being, Happiness, and Postraumatic Stress Level Scales.

Participants randomly allocated to the control group will be instructed to complete the questionnaires at baseline and follow-up but will not take part in any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Nursing students who have lived through the earthquake

Exclusion Criteria:

* Chronic respiration conditions; Heart conditions

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
1. Well-being | Baseline (Day 1) and End of Intervention (Day 2)
  The WHO-5 Well-being Index (WHO-5; World Health Organization, 1998), a widely used and validated measure, was administered pre- and post-intervention as a self-report well-being measure. Eser et al. validated and established the reliability of the WHO-5 Turkish scale in their 2019 study. Based on guidance from Eser et al. (2019), the WHO-5 Turkish scale could be used without seeking explicit permission, provided it was cited appropriately. The scale consists of five items (e.g. 'In the last 2 weeks, I have felt cheerful and in good spirits') rated on a 6-point Likert scale grading; At no time = 0, some of the time = 1, less than half of time = 2, more than half of time = 3, most of the time = 4, all of the time = 5. The scoring of the scale is done by summing the score obtained from each item, and the highest score that can be obtained from the scale is 25 and the lowest score is 0.
2. Happiness: | Baseline (Day 1) and End of Intervention (Day 2)
  The Oxford Happiness Questionnaire (OHQ-8) is an abbreviated version of the OHQ-29. It was developed to measure personal happiness and subjective well-being. The original OHQ-29 followed the format of the Beck Depression Inventory, with 20 items reversed and nine additional items added to cover aspects of happiness. The OHQ-29 is a single-scale questionnaire that can be answered on a standard six-point Likert scale. Almost half of the items (14) are negatively worded to reduce respondent bias.
3. Post-traumatic stress : | Baseline (Day 1) and End of Intervention (Day 2)
  The National Stressful Events Survey for PTSD Short Scale (NSESSS-PTSD) was used to assess PTSD symptoms. This scale is a 9-item assessment of the dimensions of post-traumatic stress disorder by DSM-5 criteria. Participants rate each item on a five-point Likert scale ranging from 0 ('never') to 4 ('always'). The total score ranges from 0 to 36, with higher scores indicating more severe symptoms of PTSD. The Turkish version of the PTSD short scale is a valid and reliable measure (alpha = 0.87) for the assessment of PTSD symptoms in the Turkish population.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided